CLINICAL TRIAL: NCT04731337
Title: Canine Occlusal Relationship Changes After Full Mouth Rehabilitation and Stainless-Steel Crown Placement Under General Anesthesia in Group of Egyptian Children; Part 1: "Before and After Study".
Brief Title: Canine Occlusal Relationship Changes After Stainless-Steel Crown Placement Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Olaya Amr Moustafa Ez ElArab ElBahnacy, Principal Investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 14422019452661
Record Dates: First submitted 2021-01-24; First posted 2021-01-29 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Full Mouth Rehabilitation; Canine Overlap Relation; General Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient's normal canine occlusal relationship (Active Comparator): The distance between the gingival zenith from the upper to the lower deciduous canines was determined by the digital calliper in millimetres (Shenzhen Jiabaili Electronic Commerce Co., Ltd) (fig1,2,3) at the right and left sides and a digital camera photographed the reading (iPhone 11 dual 12 MP Ultra-Wide and wide camera, Apple Inc.).
  Interventions: Device: Digital Caliper (Shenzhen Jiabaili Electronic Commerce Co., Ltd)
- Canine occlusal relationship after full mouth rehabilitation (Sham Comparator): The distance between the gingival zenith from the upper to the lower deciduous canines was determined by the digital calliper in millimetres (Shenzhen Jiabaili Electronic Commerce Co., Ltd) (fig1,2,3) at the right and left sides and a digital camera photographed the reading (iPhone 11 dual 12 MP Ultra-Wide and wide camera, Apple Inc.).
  Interventions: Device: Digital Caliper (Shenzhen Jiabaili Electronic Commerce Co., Ltd)

INTERVENTIONS:
Device: Digital Caliper (Shenzhen Jiabaili Electronic Commerce Co., Ltd) — Measuring the vertical distance between the tip of the upper and lower canine teeth.

SUMMARY:
The aim of the study is to Assess and compare canine occlusal relation in children with carious primary molars before they are treated by stainless steel crowns under general anaesthesia and after their placement, evaluate the possibility and the time required for the post-operative canine relation to resolve and how the treatment affects frequency and type of food intake.

DETAILED DESCRIPTION:
1. The vertical overlap was determined after closing both arches in maximum intercuspation, intruding the tongue inwards away from the occlusal surfaces.
2. After The patient had been anaesthetised, the measured values were recorded preoperatively and immediately after the treatment while the patient was unconscious.
3. In order to achieve the maximum intercuspal position (MIP) at centric occlusion, it is recommended to gently push the tongue while using a metal spatula to close the patient's mouth.
4. The distance between the gingival zenith from the upper to the lower deciduous canines was determined by the digital calliper in millimetres (Shenzhen Jiabaili Electronic Commerce Co., Ltd) at the right and left sides and a digital camera photographed the reading (iPhone 11 dual 12 MP Ultra-Wide and wide camera, Apple Inc.).
5. The tooth is anesthetised, demineralised dentine will be removed, and if a pulpotomy or pulpectomy is needed (pulpotomy with Zinconol; Dentsply Sirona, Charlotte, NC, USA) and the subsequent restoration is with high-viscosity glass ionomer cement (GIC), The tooth will be prepared by occlusal, proximal reduction and; an SCC (3M™ ESPE™ Stainless Steel Primary Molar Crowns) will be tried and adjusted to fit the tooth. The size of the PMC that is tight enough to give a feeling of 'spring back' during seating should be selected. Occlusion is checked, and the SSC will be sealed with a GIC (CVI Fuji Plus; GC).
6. Pre-operative determination of the vertical overlap of the upper and lower primary canines was done; after placement during the operation, four weeks, 2, and 6-month follow-up period.
7. Tooth preparation was done according to the principles of Spedding *1 to have 1-mm clearance between the respective tooth and the opposing tooth, and SSCs (3M ESPE, St. Paul, MN, USA) were seated, and then the operator checked occlusion.
8. After discharging the patient from the recovery room and re-establishment the function of the facial muscles, a questionnaire was taken from the parent assessing the preoperative state of the patient regarding pain and discomfort, swelling and type and frequency of food intake.
9. As part of the measurement process, a single individual was responsible for capturing the readings while another person was documenting the results with a camera. This protocol was established to ensure accuracy and consistency in the results obtained and maintain a clear measurement record.
10. Relief of symptoms and improvement of type and frequency of food intake were assessed by asking the parents.

ELIGIBILITY:
Inclusion Criteria:

1. Medical history: Normal healthy Egyptian children with no physical or mental disorders.
2. Gender: No sex predilection.
3. Age: Children from (2 to 6) years old show uncooperative behaviour.
4. Teeth: Carious teeth requiring oral dental rehabilitation under general requiring SSCs placement for primary molars.
5. Canine relationship class Ⅰ.

Exclusion Criteria:

1. Children with special health care needs or with systemic conditions.
2. Decayed primary canines with severe caries involving more than one-third of the incisal and palatal surfaces, class IV or V, crowns being built up or any incisal edge involvement.
3. Erupted permanent first molar.
4. Malocclusion i.e., Cross bite, Open bite.
5. Canine relation class Ⅱ, and Ⅲ
6. Parafunctional habits.
7. Refusal of participation.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 178 (Actual)
Dates: Start 2021-07-03 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in the canine occlusal relationship | Immediately
  The change in the canine occlusal relationship in millimeters using digital caliper
Change in the canine occlusal relationship | 4 weeks
  The change in the canine occlusal relationship in millimeters using digital caliper
Change in the canine occlusal relationship | 2 months
  The change in the canine occlusal relationship in millimeters using digital caliper
Change in the canine occlusal relationship | 6 months
  The change in the canine occlusal relationship in millimeters using digital caliper

SECONDARY OUTCOMES:
The time needed for the bite to re-adapt | "4 weeks"
  The time needed for the bite to re-adapt using digital caliper throughout days.
The time needed for the bite to re-adapt | "2 months"
  The time needed for the bite to re-adapt using digital caliper throughout days.
The time needed for the bite to re-adapt | "6 months"
  The time needed for the bite to re-adapt using digital caliper throughout days.
Child's proper masticatory function and discomfort | 4 weeks
  Child proper masticatory function and discomfort by questioning the parents.
Child proper masticatory function and discomfort | 2 months
  Child proper masticatory function and discomfort by questioning the parents.
Child proper masticatory function and discomfort | 6 months
  Child proper masticatory function and discomfort by questioning the parents.

CONTACTS AND LOCATIONS:
Overall Officials: Passant Nagi, PhD, Study Director — Passant.nagi@dentistry.cu.edu.eg
Locations (1):
- Faculty of dentistry-Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No